CLINICAL TRIAL: NCT02901353
Title: A Prospective, Single-arm, Multi-centre, Observational, Real World Registry to Evaluate Safety and Performance of the BioMime™ Morph Sirolimus Eluting Coronary Stent System for Very Long Coronary Lesions.
Brief Title: A Prospective, Single-arm, Multi-centre, Observational, Real World Registry
Acronym: Morpheus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO/MOR-I
Record Dates: First submitted 2016-08-11; First posted 2016-09-15 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sirolimus Eluting Coronary Stent System — Patient with Angina Pectoris will be enrolled for the intervention

SUMMARY:
A prospective, single-arm, multi-centre, observational, real world registry to evaluate safety and performance of the BioMime™ Morph Sirolimus Eluting Coronary Stent System for very long coronary lesions.

DETAILED DESCRIPTION:
Title:

A prospective, single-arm, multi-centre, observational, real world registry to evaluate safety and performance of the BioMime™ Morph Sirolimus Eluting Coronary Stent System for very long coronary lesions.

Short Title:

Morpheus - Global Registry Sponsor: Meril Life Sciences Pvt. Ltd

Device Used:BioMime™ Morph Sirolimus Eluting Coronary Stent System

Study population:

The utilization of the BioMime™ Morph Sirolimus Eluting Coronary Stent System implantation in very long (length ≤ 56 mm) coronary lesions in native coronary arteries with reference vessel diameter of 2.25 mm to 3.50 mm.

Enrolment:Minimum 400 patients will be enrolled

Clinical Sites:Minimum 15 sites

Objectives:Purpose of this Registry is to evaluate safety and performance of the BioMime™ Morph Sirolimus Eluting Coronary Stent System in very long (length ≤ 56 mm) coronary lesions in native coronary arteries with reference vessel diameter of 2.25 mm to 3.50 mm.

Study Design:This is a prospective, single-arm, multi-centre, observational, real world registry. All patients will be followed for up to 24 months.

Primary Outcome Measures:Freedom of target lesion failure (TLF) at 6 month and up to 24 month TLF is defined as a composite of cardiac death, myocardial infarction and target lesion revascularization.

Secondary Outcome Measures:

1. MACE at 1, 6, 12 and 24 month Defined as a composite of cardiac death, myocardial infarction attributed to the target vessel or Ischemia-driven TLR .
2. Target vessel failure at 1, 6, 12 and 24 month Defined as cardiac death, myocardial infarction attributed to the target vessel, or target vessel revascularization.
3. Academic Research Consortium (ARC) defined stent thrombosis at 1, 6, 12 and 24 months.

Definite, probable and possible stent thrombosis during acute, subacute, late and very late phase.

Other Outcome Measures:

1. Procedure Success:

   It is defined as angiographic evidence of <30% final residual stenosis of the target lesion after stent placement and no occurrence of a procedure related MACE prior to hospital discharge (for subjects with more than one lesion stented, the worse case is counted)
2. Device Success:

It is defined as angiographic evidence of <30% final residual stenosis of the target lesion using only the assigned device

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age.
2. Significant native coronary artery stenosis (> 50% by visual estimate) with lesion length of ≤56mm.
3. The patient or guardian agrees to the protocol requirements and the schedule of follow-up and provides informed written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site -

Exclusion Criteria:

1. Patients contraindicated to any of the following medications: aspirin, heparin, clopidogrel, cobalt-chromium, contrast agents and sirolimus.
2. An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 6 months post enrolment.
3. Patients who are actively participating in another drug or device investigational study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The utilization of the BioMime™ Morph Sirolimus Eluting Coronary Stent System implantation in very long (length ≤ 56 mm) coronary lesions in native coronary arteries with reference vessel diameter of 2.25 mm to 3.50 mm.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Freedom of target lesion failure | TLF at 6 month
  composite of cardiac death, myocardial infarction and target lesion revascularization.
Freedom of target lesion failure | TLF upto 24 months
  composite of cardiac death, myocardial infarction and target lesion revascularization.

SECONDARY OUTCOMES:
MACE | 1, 6, 12 and 24 month
  composite of cardiac death, myocardial infarction attributed to the target vessel or Ischemia-driven TLR.
Target vessel failure | 1, 6, 12 and 24 month
  cardiac death, myocardial infarction attributed to the target vessel, or target vessel revascularization.
Academic Research Consortium (ARC) defined stent thrombosis | 1, 6, 12 and 24 month
  Definite, probable and possible stent thrombosis during acute, subacute, late and very late phase.

OTHER OUTCOMES:
Procedure Success | Before Discharge
  Angiographic evidence of <30% final residual stenosis of the target lesion after stent placement and no occurrence of a procedure related MACE prior to hospital discharge (for subjects with more than one lesion stented, the worse case is counted)
Device Success | Before Discharge
  Angiographic evidence of <30% final residual stenosis of the target lesion using only the assigned device

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Bela Merkely, MD, Ph.D, D.Sc, Principal Investigator — University of Semmelweis; Dr. Szűk Tibor, Ph.D, MD, Principal Investigator — University of Debrecen; Dr. P. Agostoni, Ph.D, MD, Principal Investigator — St. Antonius Nieuwegein; Dr. Imad A Haddad, MD, Principal Investigator — Jordan Hospital; Dr. Ramesh Singh, MBBS, MRCP, Principal Investigator — University Malaya Medical Centre (UMMC)
Locations (5):
- Hungary (2):
  - University of Semmelweis, Budapest, Europe
  - University of Debrecen, Debrecen, Europe
- Jordan Hospital, Amman, Jordan
- University Malaya Medical Centre (UMMC), Kuala Lumpur, Selangor, Malaysia
- St. Antonius Hospital, Nieuwegein, Germany, Netherlands

IPD SHARING:
Plan to Share IPD: No